CLINICAL TRIAL: NCT00309452
Title: Randomized Trial of Usual Care Versus Specialized, Phase-specific Care in the Public Sector for First Episode Psychosis.
Brief Title: Specialized Treatment Early in Psychosis (STEP)
Acronym: STEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0601001013
Record Dates: First submitted 2006-03-29; First posted 2006-03-31 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2016-12

CONDITIONS: Schizophrenia and Disorders With Psychotic Features
Keywords: First episode psychosis; Specialized care; Phase-specific treatment; Schizophrenia; Disorders with psychotic features
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders; Schizophrenia | interventions — Cognitive Remediation; Dosage Forms; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment as usual (Active Comparator): Referral to community providers.
  Interventions: Other: Treatment as Usual in the community
- STEP Care (Experimental): Integrated and comprehensive treatment provided by a specialized team in a public mental health center.Interventions include pharmacotherapy, family education, cognitive behavioral group and individual psychotherapy and case management focused on vocational rehabilitation.
  Interventions: Behavioral: Cognitive Behavioral Group Therapy; Behavioral: Cognitive remediation; Drug: Medications; Behavioral: MFG; Behavioral: Assertive case management

INTERVENTIONS:
Behavioral: Cognitive Behavioral Group Therapy — once per week
  Arms: STEP Care
Behavioral: Cognitive remediation — as needed
  Arms: STEP Care
Drug: Medications — Individualized prescription of psychotropic medications including but not restricted to antipsychotic, antidepressant and mood stabilizers.
  Arms: STEP Care
Behavioral: MFG — Multi-Family psychoeducation Group based on the model published by McFarlane et al.
  Arms: STEP Care
Behavioral: Assertive case management — Meetings with an individual clinician (social work or nursing) who provides supportive psychotherapy, helps assist with vocational and educational supports.
  Arms: STEP Care
Other: Treatment as Usual in the community — Subjects randomized to this arm either return to their existing outpatient psychiatrist or, if they do not have one yet, are referred by the clinic to preferred providers in the community. The nature of the interventions provided is variable and is being monitored by the research clinic.
  Arms: Treatment as usual

SUMMARY:
The purpose of this study is to understand the effectiveness of a specialized package of phase-specific treatments for individuals in the midst of their first episode of psychosis. The pharmacologic and psychosocial treatments will be delivered within a state public mental health center.

DETAILED DESCRIPTION:
We propose to conduct a clinical trial for first episode psychosis patients not eligible for CMHC services that will compare randomized access to care at CMHC versus the usual procedure of referral to community providers outside CMHC. Patients randomized to access to CMHC services will receive multifaceted, intensive, phase-specific care delivered by a specialized clinical team. This care will include five principal components: antipsychotic prescription, multi-family group therapy, group cognitive behavioral therapy, cognitive remediation and individual case management including supportive, problem solving approaches and a focus on resumption of movement towards educational and/or employment related goals. All consenting subjects will undergo research evaluations every six months for up to five years. Outcomes will be assessed in the domains of re-admission (primary outcome), relapse, symptoms, overall functioning, quality of life, education and employment, treatment satisfaction, adherence, substance use, adverse events (including self-harm) and economic measures including service use, cost of care and forensic data.

ELIGIBILITY:
Inclusion Criteria:

1. Age 16-45
2. Meets DSM-IV schizophrenia spectrum psychosis or affective psychosis according to the SCID
3. ≤8 weeks of received antipsychotic treatment lifetime at time of referral
4. Willing to be treated in New Haven

Exclusion Criteria:

1. Psychosis believed due to substance use (based on the SCID)
2. Unable or unwilling to give informed consent
3. MR as indicated by receipt of services from Dept of Mental Retardation

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2006-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vinod H Srihari, M.D., Principal Investigator — Yale University School of Medicine & Connecticut Mental Health Center; Scott Woods, M.D., Study Chair — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

REFERENCES:
- [Background] Srihari VH, Breitborde NJ, Pollard J, Tek C, Hyman L, Frisman LK, McGlashan TH, Jacobs S, Woods SW. Public-academic partnerships: early intervention for psychotic disorders in a community mental health center. Psychiatr Serv. 2009 Nov;60(11):1426-8. doi: 10.1176/appi.ps.60.11.1426. PMID 19880454
- [Background] Breitborde NJ, Woods SW, Srihari VH. Multifamily psychoeducation for first-episode psychosis: a cost-effectiveness analysis. Psychiatr Serv. 2009 Nov;60(11):1477-83. doi: 10.1176/ps.2009.60.11.1477. PMID 19880465
- [Background] Breitborde NJ, Srihari VH, Pollard JM, Addington DN, Woods SW. Mediators and moderators in early intervention research. Early Interv Psychiatry. 2010 May;4(2):143-52. doi: 10.1111/j.1751-7893.2010.00177.x. PMID 20536970
- [Background] Saksa JR, Cohen SJ, Srihari VH, Woods SW. Cognitive behavior therapy for early psychosis: a comprehensive review of individual vs. group treatment studies. Int J Group Psychother. 2009 Jul;59(3):357-83. doi: 10.1521/ijgp.2009.59.3.357. PMID 19548785
- [Background] Breitborde NJ, Srihari VH, Woods SW. Review of the operational definition for first-episode psychosis. Early Interv Psychiatry. 2009 Nov;3(4):259-65. doi: 10.1111/j.1751-7893.2009.00148.x. PMID 22642728
- [Background] Srihari VH, Shah J, Keshavan MS. Is early intervention for psychosis feasible and effective? Psychiatr Clin North Am. 2012 Sep;35(3):613-31. doi: 10.1016/j.psc.2012.06.004. Epub 2012 Jul 21. PMID 22929869
- [Background] Ozkan B, Phutane V, Jonas E, Tek C, Srihari V. Hoofbeats and zebras: neurodegenerative disorder presenting as a "first episode" of psychosis. Gen Hosp Psychiatry. 2011 Jul-Aug;33(4):412.e1-3. doi: 10.1016/j.genhosppsych.2011.03.011. Epub 2011 May 5. PMID 21762843
- [Result] Dodds TJ, Phutane VH, Stevens BJ, Woods SW, Sernyak MJ, Srihari VH. Who is paying the price? Loss of health insurance coverage early in psychosis. Psychiatr Serv. 2011 Aug;62(8):878-81. doi: 10.1176/ps.62.8.pss6208_0878. PMID 21807825
- [Result] Perez VB, Ford JM, Roach BJ, Woods SW, McGlashan TH, Srihari VH, Loewy RL, Vinogradov S, Mathalon DH. Error monitoring dysfunction across the illness course of schizophrenia. J Abnorm Psychol. 2012 May;121(2):372-87. doi: 10.1037/a0025487. Epub 2011 Nov 7. PMID 22060947
- [Result] Breitborde NJ, Kleinlein P, Srihari VH. Self-determination and first-episode psychosis: associations with symptomatology, social and vocational functioning, and quality of life. Schizophr Res. 2012 May;137(1-3):132-6. doi: 10.1016/j.schres.2012.02.026. Epub 2012 Mar 22. PMID 22445463
- [Result] Phutane VH, Tek C, Chwastiak L, Ratliff JC, Ozyuksel B, Woods SW, Srihari VH. Cardiovascular risk in a first-episode psychosis sample: a 'critical period' for prevention? Schizophr Res. 2011 Apr;127(1-3):257-61. doi: 10.1016/j.schres.2010.12.008. Epub 2011 Jan 15. PMID 21242060
- [Result] Srihari VH, Tek C, Kucukgoncu S, Phutane VH, Breitborde NJ, Pollard J, Ozkan B, Saksa J, Walsh BC, Woods SW. First-Episode Services for Psychotic Disorders in the U.S. Public Sector: A Pragmatic Randomized Controlled Trial. Psychiatr Serv. 2015 Jul;66(7):705-12. doi: 10.1176/appi.ps.201400236. Epub 2015 Feb 2. PMID 25639994
- See also: Related Info — http://www.step.yale.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 512 requests for information, of which 491 were screened by phone for eligibility. 284 were excluded. Of the 207 who completed a full in-person eligibility assessment, 2 were deemed ineligible and 29 were provided STEP care without randomization in an initial pilot (data not included). 120 of the remaining 176 patients were enrolled.
Period: Overall Study
Arm/Group | Treatment as Usual | STEP Care
Started | 60 | 60
Completed | 57 | 60
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment as Usual | STEP Care | Total
Number analyzed (Participants) | 57 | 60 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.6 (5.3) | 22.4 (4.5) | 22.5 (4.9)
Gender [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 46 | 49 | 95
Global Assessment of Functioning [Mean (Standard Deviation); unit: units on a scale] — The Global Assessment of Functioning (GAF) is a numeric scale (1 through 100) used by mental health clinicians and physicians to rate subjectively the social, occupational, and psychological functioning of adults, e.g., how well or adaptively one is meeting various problems-in-living. The higher the score, the better functioning the subject.
  units on a scale | 34.42 (10.43) | 36.22 (12.89) | 35.88 (13.04)
PANNS Positive and Negative Symptom Scale [Mean (Standard Deviation); unit: units on a scale] — The Positive scale has7 Items, (minimum score = 7, maximum score = 49). With a higher score indicates more severe symptoms.
  The Negative scale has 7 Items, (minimum score = 7, maximum score = 49). With a higher score indicates more severe symptoms.
  The General Psychopathology scale has 16 Items, (minimum score = 16, maximum score = 112). With a higher score indicates more severe symptoms.
  The range for the PANSS Total score is minimum = 30, maximum = 210. With a higher score indicates more severe symptoms.
  units on a scale
    Positive Dimension | 19.60 (5.90) | 20.75 (6.74) | 20.21 (6.36)
    Negative Dimension | 17.01 (5.40) | 17.82 (6.42) | 17.44 (5.95)
    General Symptoms | 33.70 (8.56) | 33.42 (8.62) | 33.56 (8.56)
    Total | 70.33 (15.52) | 72.0 (16.76) | 71.21 (16.14)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Hospitalized
Time Frame: 1 year after enrollment
Measure: Number; unit: participants
Arm/Group | Treatment as Usual | STEP Care
Number analyzed (Participants) | 57 | 60
participants | 25 | 14
Statistical Analysis 1: Comparison: Treatment as Usual vs STEP Care; Between groups comparison for hospitalization rates, adjusted for pretreatment hospitalization; Test type: Superiority or Other; p = 0.018, Chi-squared, Corrected

2. Secondary Outcome: Relapse
Description: Data was not collected, instead Hospitalization (primary outcome) was used as a proxy
Time Frame: every 6 months
Arm/Group | Treatment as Usual | STEP Care
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Overall Functioning- Global Assessment of Functioning
Description: The Global Assessment of Functioning (GAF) is a numeric scale (1 through 100) used by mental health clinicians and physicians to rate subjectively the social, occupational, and psychological functioning of adults, e.g., how well or adaptively one is meeting various problems-in-living. A higher score indicates better functioning.
  The score reported is a change from baseline. The change was calculated as score at 12 months minus score from baseline. A positive score indicates higher functioning.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment as Usual | STEP Care
Number analyzed (Participants) | 57 | 60
units on a scale
  Baseline | 34.42 (10.43) | 36.22 (12.89)
  Change from baseline | 20.38 (16.61) | 22.22 (15.46)

4. Secondary Outcome: Quality of Life- Heinrich's Quality of Life Scale
Description: The Quality of Life Scale (QLS) is a 21-item scale rated from a semistructured interview providing information on symptoms and functioning during the preceding 4 weeks. Each item is rated on a seven point scale, and a higher score reflects normal or unimpaired functioning. The range is from 0 to 126.
  The score reflected is a change from baseline. Total score at 12 months minus total score at baseline. A positive score indicates better mental health.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment as Usual | STEP Care
Number analyzed (Participants) | 57 | 60
units on a scale
  Baseline | 59.45 (18.02) | 59.87 (22.25)
  Change from Baseline | -.80 (20.18) | 9.81 (29.85)

5. Secondary Outcome: Vocationally Engaged
Time Frame: 1 year after enrollment
Population: 20 subjects from the treatment as usual arm were lost to follow-up. 12 subjects from STEP Care arm were lost to follow up.
Measure: Number; unit: participants
Arm/Group | Treatment as Usual | STEP Care
Number analyzed (Participants) | 37 | 48
participants | 26 | 44
Statistical Analysis 1: Comparison: Treatment as Usual vs STEP Care; Between groups comparison for vocational engagement, adjusted for pretreatment vocational engagement; Test type: Superiority or Other; p = 0.002, Chi-squared, Corrected

6. Secondary Outcome: Treatment Satisfaction
Time Frame: every 6 months
Population: Data was not collected
Arm/Group | Treatment as Usual | STEP Care
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Adherence- in Contact With Mental Health Services
Description: Number of participants in contact with mental health services. Collected via self-report.
Time Frame: 1 year
Population: Patients were lost to follow up. 15 subjects in the Treatment as Usual arm, and 15 subjects in the STEP care arm.
Measure: Number; unit: participants
Arm/Group | Treatment as Usual | STEP Care
Number analyzed (Participants) | 42 | 45
participants | 33 | 39

8. Secondary Outcome: Substance Use
Time Frame: every 6 months
Population: This was not a planned primary or secondary outcome in our analysis (though collected at baseline) and because of significant attrition we did not report on this outcome despite having phone call f/u data on other outcomes. We did not believe phone reports on this outcome would produce reliable data.
Arm/Group | Treatment as Usual | STEP Care
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Subjects Who Committed Self-harm and Violence
Description: The number of subjects who committed an act of self-harm or violence. This data was collected at 12 months.
Time Frame: 12 months
Population: This data was collected, numbers reflect actual data.
Measure: Number; unit: participants
Arm/Group | Treatment as Usual | STEP Care
Number analyzed (Participants) | 57 | 60
participants | 0 | 0

10. Secondary Outcome: Medication (Including Metabolic) Side Effects
Time Frame: every 6 months
Population: data no collected
Arm/Group | Treatment as Usual | STEP Care
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Economic Measures Including Service Use, Cost of Care and Forensic Data.
Description: Total annual cost per patient
Time Frame: every 6 months
Measure: Mean (Standard Error); unit: dollars
Arm/Group | Treatment as Usual | STEP Care
Number analyzed (Participants) | 57 | 60
dollars | 12157.46 (2948.83) | 7625.22 (2539.70)

ADVERSE EVENTS:
Arm/Group | Treatment as Usual | STEP Care
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/60
Other Adverse Events (participants affected / at risk) | 0/57 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No